CLINICAL TRIAL: NCT04788069
Title: Effect of Sourdough Breads Consumption on Postprandial Responses, Satiety and Food Intake at Subsequent Meal
Acronym: SUPPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: S64824
Record Dates: First submitted 2021-02-24; First posted 2021-03-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Energy Intake; Appetite Regulation
MeSH Terms: interventions — Bread

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wholemeal bread (Active Comparator): Treatment with wholemeal bread
  Interventions: Dietary Supplement: Wholemeal bread
- Sourdough bread (Active Comparator): Treatment with sourdough bread
  Interventions: Dietary Supplement: Sourdough bread
- Bread with sourdough (Active Comparator): Treatment with bread with sourdough
  Interventions: Dietary Supplement: Bread with sourdough

INTERVENTIONS:
Dietary Supplement: Wholemeal bread — 180g wholemeal bread/day + fixed portion at test day
  Arms: Wholemeal bread
Dietary Supplement: Sourdough bread — 180g sourdough bread/day + fixed portion at test day
  Arms: Sourdough bread
Dietary Supplement: Bread with sourdough — 180g bread with sourdough/day + fixed portion at test day
  Arms: Bread with sourdough

SUMMARY:
During this project the effect of different types of sourdough breads consumption on satiety, energy intake at subsequent meal and postprandial metabolic responses, will be investigated.

DETAILED DESCRIPTION:
A 3-phase randomised cross-over trial will be applied consisting of 3 intervention periods of 2 weeks, with a test day performed at the last day of each intervention period. During each intervention period, participants will consume a fixed amount of test bread, replacing their regular bread, and they will keep food and stool diaries preceding each Test-day. Faecal samples will be collected before each Test-day. On the Test-day, participants will perform a gastric emptying breath test. Furthermore, blood samples and appetite ratings will be collected at regular time points after consumption of the test bread for measurement of glucose, insulin, gut peptides, short-chain fatty acids (SCFA) and blood lipids. Food intake will be assessed by offering the subjects a standard lunch to be consumed ad-libitum.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants
* age range 18 - 50
* BMI range 18.5 - 25.0 kg/m2 at screening visit
* Regular eating pattern (3 meals per day on at least 5 days per week)
* Willingness to consume bread (180 g) on a daily base
* Stable body weight for the last 6 months

Exclusion Criteria:

* Currently smoking (has smoked in the last 28 days) or willingness to smoke during the study period
* Pregnancy, lactation or wish to become pregnant during the study period
* Family history of diabetes
* Previous or current gastrointestinal or endocrine disorders
* Previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)
* Intake of prescription medication
* Coeliac disease or gluten sensitivity
* Use of pre- or probiotics within one month preceding the study
* Use of antibiotics within 3 months preceding the study
* Excessive concern about eating habits or body weight as evidenced from scores < 18 on the restraint and disinhibition subscales of the Three-Factor Eating Questionnaire (Stunkard & Messick, 1985)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Appetite measurements | During test day 1 (up to 4 hours)
  Appetite in response to test meal, will be measured using 100 millimeter (mm) Visual Analogue Scales (VAS) before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Appetite measurements | During test day 2 (up to 4 hours)
  Appetite in response to test meal, will be measured using 100 millimeter (mm) Visual Analogue Scales (VAS) before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Appetite measurements | During test day 3 (up to 4 hours)
  Appetite in response to test meal, will be measured using 100 millimeter (mm) Visual Analogue Scales (VAS) before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Food intake at subsequent meal | During test day 1 (240 minutes after ingestion of breakfast)
  Weighted amounts of ad-libitum food offered minus the weighted leftovers
Food intake at subsequent meal | During test day 2 (240 minutes after ingestion of breakfast)
  Weighted amounts of ad-libitum food offered minus the weighted leftovers
Food intake at subsequent meal | During test day 3 (240 minutes after ingestion of breakfast)
  Weighted amounts of ad-libitum food offered minus the weighted leftovers

SECONDARY OUTCOMES:
Oral processing behaviour | During test day 1 (up to 15 minutes)
  Participants will be video-recorded to measure oral processing behaviour of the test meal
Oral processing behaviour | During test day 2 (up to 15 minutes)
  Participants will be video-recorded to measure oral processing behaviour of the test meal
Oral processing behaviour | During test day 3 (up to 15 minutes)
  Participants will be video-recorded to measure oral processing behaviour of the test meal
Blood lipids | During test day 1
  Plasma total cholesterol, triglycerides, LDL and HDL cholesterol, colourimetrically
Blood lipids | During test day 2
  Plasma total cholesterol, triglycerides, LDL and HDL cholesterol, colourimetrically
Blood lipids | During test day 3
  Plasma total cholesterol, triglycerides, LDL and HDL cholesterol, colourimetrically
Glucose response | During test day 1 (up to 4 hours)
  Blood glucose response will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes)
Glucose response | During test day 2 (up to 4 hours)
  Blood glucose response will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes)
Glucose response | During test day 3 (up to 4 hours)
  Blood glucose response will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes)
Insulin response | During test day 1 (up to 4 hours)
  Blood C-peptide (as indicator of insulin response) will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes).
Insulin response | During test day 2 (up to 4 hours)
  Blood C-peptide (as indicator of insulin response) will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes).
Insulin response | During test day 3 (up to 4 hours)
  Blood C-peptide (as indicator of insulin response) will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes).
Incretin hormones | During test day 1 (up to 4 hours)
  Incretin hormones (GLP-1 and PYY) will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes).
Incretin hormones | During test day 2 (up to 4 hours)
  Incretin hormones (GLP-1 and PYY) will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes).
Incretin hormones | During test day 3 (up to 4 hours)
  Incretin hormones (GLP-1 and PYY) will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240 minutes).
Short-chain-fatty-acids | During test day 1 (up to 8 hours)
  Short-chain-fatty-acids will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, 480 minutes).
Short-chain-fatty-acids | During test day 2 (up to 8 hours)
  Short-chain-fatty-acids will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, 480 minutes).
Short-chain-fatty-acids | During test day 3 (up to 8 hours)
  Short-chain-fatty-acids will be measured through blood samples collected via placed catheter before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, 480 minutes).
Short-chain-fatty-acids | 1 time after intervention with each bread type (totally 3 times over a period of 10 weeks)
  Faecal (GC-FID)
Gastric emptying rate | During test day 1 (up to 4 hours)
  Gastric emptying rate will be measured through 13C-octanoic acid breath samples collected before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Gastric emptying rate | During test day 2 (up to 4 hours)
  Gastric emptying rate will be measured through 13C-octanoic acid breath samples collected before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Gastric emptying rate | During test day 3 (up to 4 hours)
  Gastric emptying rate will be measured through 13C-octanoic acid breath samples collected before eating (i.e. 0 minute) and at respective time points after completion of test meal (I.e. 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes).
Free-living energy intake | 4 days during intervention with each bread type (totally 3x4 days over a period of 10 weeks)
  4-day food diaries, mobile app
Stool shape and consistency | 4 days during intervention with each bread type (totally 3x4 days over a period of 10 weeks)
  4-day stool diaries, the Bristol Stool Score
Change in Gut microbiota composition | 1 time after intervention with each bread type (totally 3 times over a period of 10 weeks)
  Change in Gut microbiota composition after consumption of each test meal for 14 days will be analysed using the relative abundance of bacterial taxa according to 16S rRNA sequencing data

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Prof., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven/ UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No